CLINICAL TRIAL: NCT07101315
Title: Early Versus Delayed Laparoscopic Cholecystectomy for Acute Cholecystitis: A Prospective Study Adjusting for Confounding by Indication
Brief Title: Early Versus Delayed Laparoscopic Cholecystectomy for Acute Cholecystitis
Acronym: EDLC-AC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sana'a University (Other)
Collaborators: Al-Thawra Modern General Hospital (Other); Al-Kuwait University Hospital (Unknown)
Responsible Party: Principal Investigator, Haitham Mohammed Jowah, Lecturer, Sana'a University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SanaaU-Chole-001
Record Dates: First submitted 2025-07-27; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Acute Cholecystitis
Keywords: Laparoscopic Cholecystectomy; Gallstones; Biliary Disease; Surgical Timing
MeSH Terms: conditions — Cholecystitis, Acute; Gallstones; Gallbladder Diseases | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Laparoscopic Cholecystectomy (ELC) (Experimental): Participants underwent laparoscopic cholecystectomy within 72 hours of symptom onset during the index hospital admission.
  Interventions: Procedure: Laparoscopic Cholecystectomy
- Delayed Laparoscopic Cholecystectomy (DLC) (Active Comparator): Participants received initial non-operative management with antibiotics and analgesics, followed by elective laparoscopic cholecystectomy 6-8 weeks later.
  Interventions: Procedure: Laparoscopic Cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic Cholecystectomy — Standard four-port laparoscopic cholecystectomy was performed by a specialist or resident surgeon.

SUMMARY:
The goal of this clinical trial is to learn if performing gallbladder surgery early is as safe and effective as delaying it for people with acute cholecystitis (a sudden gallbladder infection). The main questions it aims to answer are:

* Do participants who have early surgery have a similar rate of complications compared to those who have delayed surgery?
* How does the timing of surgery affect the length of the hospital stay?

Researchers will compare two groups:

1. An early surgery group
2. A delayed surgery group

Participants in the early surgery group had their gallbladder removed within 72 hours of when their symptoms started. Participants in the delayed surgery group were first treated with medications and had their surgery 6-8 weeks later.

ELIGIBILITY:
Inclusion Criteria:

* Yemeni nationals aged 18-70 years
* A clinical diagnosis of acute cholecystitis confirmed by clinical presentation, laboratory findings, and imaging studies
* Symptom duration of less than 72 hours at presentation
* Fitness for general anesthesia (American Society of Anesthesiologists [ASA] physical status classification I-III)
* Provision of written informed consent

Exclusion Criteria:

* Evidence of choledocholithiasis or acute cholangitis
* Severe comorbidities precluding surgery (ASA class IV-V)
* Coagulopathy (INR >1.5 or platelet count <100,000/μL)
* Pregnancy
* Previous major upper abdominal surgery
* Patient refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Overall Postoperative Complications | Within 30 days post-surgery
  Incidence of any postoperative complication within 30 days
Conversion to Open Surgery | Intraoperative
  Rate of conversion from laparoscopic to open cholecystectomy during the procedure.
Operative Time | Intraoperative
  Duration of surgery, measured in minutes from skin incision to skin closure.

SECONDARY OUTCOMES:
Postoperative Length of Hospital Stay | Up to 30 days post-surgery
  Number of days from surgery to hospital discharge.
Duration of Postoperative Pain | Up to 30 days post-surgery
  Number of days from surgery until the participant was free of the need for analgesic medication.
Time to Return to Normal Daily Activities | Up to 30 days post-surgery
  Number of days from surgery until the participant reported a full return to normal daily activities.
30-Day Readmission Rate | 30 days
  Rate of unplanned hospital readmission for any cause within 30 days of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Issa, Professor, Principal Investigator — Sana'a University
Locations (2):
- Yemen (2):
  - Al-Kuwait University Hospital, Sanaa
  - Al-Thawra Modern General Hospital, Sanaa

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in this article, after publication. This includes data for all primary and secondary outcome measures. The study protocol will not be shared.
Time Frame: Data will be available beginning 3 months after article publication and the access period will remain open for 5 years.
Access Criteria: Data will be made available to qualified researchers for meta-analysis or other secondary analyses consistent with the original aims of the study. Researchers must submit a methodologically sound proposal to the corresponding author at h.jowah@su.edu.ye. A signed data access agreement will be required prior to the release of any data.